CLINICAL TRIAL: NCT00667095
Title: Evaluation of the Efficacy of Botulinum-A Toxin/DMSO Instillation in the Treatment of Women With Over Active Bladder (OAB) Syndrome and/or Urinary Urge Incontinence
Brief Title: Over Active Bladder Instillation Study - Botox
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated early due to PI's extended medical leave.
Sponsor: Mayo Clinic (Other)
Responsible Party: Steven P. Petrou, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-007399
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Overactive Bladder; Urinary Urge Incontinence; Urinary Incontinence; Detrusor Hyperreflexia; Urge Incontinence
Keywords: OAB; Over Active Bladder; overactive bladder; Urinary Urge Incontinence; Urinary Incontinence; Botox; DMSO; bladder instillation; instillation; detrusor hyperreflexia; urge incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence | interventions — Botulinum Toxins, Type A; Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botox and DMSO instillation (Experimental): Botulinum-A Toxin (Botox) 300 units in 50 cubic centimeters of Dimethyl Sulfoxide (DMSO) 50% w/w aqueous solution
  Interventions: Drug: Botox Instillation; Drug: DMSO Instillation
- DMSO instillation (Placebo Comparator): Dimethyl Sulfoxide (DMSO) 50% w/w aqueous solution, 50 cubic centimeters
  Interventions: Drug: DMSO Instillation

INTERVENTIONS:
Drug: Botox Instillation — Botox instilled into the bladder via ureteral catheter and retained for up to 30 minutes then spontaneously voided.
  Other Names: Botulinum-A Toxin; Botox
  Arms: Botox and DMSO instillation
Drug: DMSO Instillation — DMSO 50% w/w aqueous solution; 50 cubic centimeters instilled into the bladder via ureteral catheter and retained up to 30 minutes then spontaneously voided.
  Other Names: Dimethyl Sulfoxide; DMSO

SUMMARY:
The purpose of this study is to determine whether women with overactive bladder (OAB) who receive direct instillation via a catheter of a Botulinum-A Toxin (Botox) with Dimethyl Sulfoxide (DMSO) solution experience significantly better improvement of their OAB symptoms when compared to a similar group of women with OAB who receive instillation of DMSO only.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of catheter-based instillation of a solution of Botox/DMSO as a novel method for treating women with overactive bladder (OAB) and secondary urinary incontinence who have failed oral pharmacologic therapy. This study will test the broad hypothesis that administration of Botox/DMSO instillations into the bladder with a urethral catheter can significantly improve symptoms and quality of life in patients with OAB when compared to DMSO installations alone. Explicitly, we hypothesize that scores on the validated Incontinence Quality of Life (I-QOL) questionnaire of women with OAB who receive Botox/DMSO instillation will be much improved at three-month follow-up compared to similar women receiving DMSO instillation alone. Our long-term goal is to offer women with detrusor hyperreflexia or OAB a less invasive alternative to surgery and an alternative to anticholinergic by mouth medications. In support of this effort, we are proposing a randomized, double-blind, placebo controlled clinical trial to be conducted in the Department of Urology at Mayo Clinic, Jacksonville, Florida.

Note: The study was terminated early in July of 2011 due to an extended medical absence of the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Female patient aged 18 years or older
* No evidence of stress urinary incontinence on physical examination or urodynamics
* Patients who have failed prior drug therapy for overactive bladder or detrusor hyperreflexia
* Patients with symptoms and signs of OAB, detrusor hyperreflexia, urinary urgency, urinary urge incontinence.
* Patient who is mentally competent with the ability to understand and comply with the requirements of the study
* Patient who agrees to be available for the follow-up evaluations as required by the protocol
* Patient who has given signed informed consent

Exclusion Criteria:

* Patient with Post-Void Residual Urine (PVRU) greater than 100 ml on repeated measures. (Patient with a single PVRU of >100 ml and followed by two consecutive PVRU measurements of <100 ml may be included in the study)
* Patient with greater than vesicoureteral reflux grade 1, interstitial cystitis, genitourinary fistulae
* Patient with pelvic organ prolapse stage III or IV, i.e. the most distal part of the prolapse protruding more than 1 cm beyond the hymen (>+1), at straining
* Patient with un-investigated hematuria
* Patient with lower tract genitourinary malignancies
* Patient on current medication for stress urinary incontinence, such as alpha-adrenergic agonists or duloxetine, within three weeks prior to completing the baseline Bladder Diary (estrogen therapy on a stable dose for at least two months prior to study start is allowed)
* Patient with ongoing complications of prior anti-incontinence surgery
* Patient who is pregnant, lactating, or planning to become pregnant within the study period
* Patient who has received pelvic radiation
* Patient with any condition, which could lead to significant postoperative complications, including current infection and uncontrolled diabetes.
* Patient who is morbidly obese (defined as BMI > 40 Kg/m2)
* Patient who is bedridden, institutionalized or in such physical condition that she cannot move to the closest bathroom without assistance from another person
* Patient with current or acute urinary tract infection, including cystitis or urethritis. (Patient with such infections should be treated with antibiotics, with subsequent urinalysis tests confirming the absence of such infection before study inclusion)
* Patient with any condition that would preclude treatment due to contraindications and/or warnings in the study product's labeling
* Patient on immunomodulatory therapy (suppressive or stimulatory)
* Patient with known lidocaine hypersensitivity or hypersensitivity to any anesthetics to be used during the treatment session/surgical procedure
* Patient with a concurrent use of another study product within two weeks prior to study start, or who concurrently participate in any other clinical study
* Any disease that in the opinion of the Investigator would make the patient unsuitable for the study
* Patient with a life expectancy of less than 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Petrou, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Petrou SP, Parker AS, Crook JE, Rogers A, Metz-Kudashick D, Thiel DD. Botulinum a toxin/dimethyl sulfoxide bladder instillations for women with refractory idiopathic detrusor overactivity: a phase 1/2 study. Mayo Clin Proc. 2009 Aug;84(8):702-6. doi: 10.4065/84.8.702. PMID 19648387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 25 subjects were recruited from 10/21/2008 to 8/19/2010. Three of these were determined to be screen failures before randomization, and another one was withdrawn prior to randomization. Twenty one subjects were randomized: 11 to Botox/DMSO, and 10 to DMSO only.
Period: Overall Study
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox and DMSO Instillation | DMSO Instillation | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 58 [36 to 85] | 71 [38 to 93] | 68 [36 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
Smoking Status [Number; unit: participants]
  Never smoked | 4 | 6 | 10
  Past smoker | 6 | 4 | 10
  Current smoker | 1 | 0 | 1
History of Hypertension [Number; unit: participants]
  Hypertension | 6 | 7 | 13
  No hypertension | 5 | 3 | 8
History of Urinary Tract Infections (UTIs) [Number; unit: participants]
  Previous history of UTIs | 10 | 10 | 20
  No previous UTIs | 1 | 0 | 1
Number of Vaginal Births [Number; unit: participants]
  0 vaginal births | 3 | 3 | 6
  1-2 vaginal births | 4 | 1 | 5
  ≥ 3 vaginal births | 4 | 6 | 10
Body Mass Index [Median (Full Range); unit: kg/m^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat. A body mass index of under 20 is considered to be underweight, while a body mass index between 20 to 25 is considered healthy. A body mass index in the range of 25 to 30 is regarded as overweight. A body mass index over 30 is regarded as obese.
  kg/m^2 | 26 [22 to 38] | 30 [19 to 40] | 27 [19 to 40]
Post-Void Residual Urine [Median (Full Range); unit: mL] | 15 [0 to 91] | 29 [0 to 116] | 17 [1 to 116]
Incontinent Episodes during 24 Hours [Median (Full Range); unit: Episodes] — The study coordinator instructed the subject to keep record of any incontinence episodes during the 24-hour period prior to their baseline visit.
  Episodes | 6 [0 to 8] | 3 [1 to 9] | 4 [0 to 9]
Median 24 Hour Pad Weight [Median (Full Range); unit: g] — Prior to the baseline visit, the study coordinator weighed standard pads provided to the subject for the study time period. The study coordinator instructed the subject to bring in any pads used during the 24-hour period prior to the baseline visit. The study coordinator recorded the 24-hour pad weight into the study dataset.
  g | 166 [0 to 585] | 179 [5 to 1618] | 166 [0 to 1618]
Median Number of Pads Per Day [Median (Full Range); unit: pads] | 4 [1 to 9] | 5 [3 to 8] | 5 [1 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Change in Incontinence Quality of Life (I-QoL) Score
Description: The I-QoL measures the effect of urinary incontinence on quality of life. It is divided into 3 subscales: 1) avoidance and limiting behavior, 2) psychosocial impact, and 3) social embarrassment. The I-QOL is comprised of 22 items, each with the response scale from '1= Extremely' to '5= Not at all'.
  A mean score for each subscale is calculated (averaging the scores for the items in each subscale) as well as a total score for all 22 items (sum of all subscale scores). The scores are then transformed to a 'Scale score' ranging from 0-100 points for ease of interpretation: Scale score = (sum of the items - lowest possible score)/possible raw score range X 100. Higher scores indicate less impact of incontinence on quality of life.
Time Frame: Baseline, 1 month, 3 months
Population: Analysis was done according to the principle of intention-to-treat. The sample size was reduced to 9 in the Dimethyl Sulfoxide (DMSO) instillation arm at 3 months due to withdrawal for reasons unrelated to study (cancer).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Number analyzed (Participants) | 11 | 10
units on a scale
  Change from baseline to 1 month | 9.6 (13.3) | -3.9 (11.6)
  Change from baseline to 3 months (n=11, 9) | 8.6 (14.4) | -4.0 (9.3)
Statistical Analysis 1: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 1 month; Test type: Superiority or Other; p = 0.024, t-test, 2 sided
Statistical Analysis 2: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 3 months; Test type: Superiority or Other; p = 0.036, t-test, 2 sided

2. Secondary Outcome: Change in Incontinence Impact Questionnaire Short Form (IIQ-7)
Description: The IIQ-7 measures the effect of urinary incontinence on quality of life. It is comprised of 7 items, each with the response scale from "0=Not at all" to "3=Greatly." The scores can range from 0 to 21; a low score indicates less impact of incontinence on quality of life.
Time Frame: baseline, 1 month, 3 months
Population: Analysis was done according to the principle of intention-to-treat. The sample size was reduced to 9 in the Dimethyl Sulfoxide (DSMO) instillation arm at 3 months due to withdrawal for reasons unrelated to study (cancer).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Number analyzed (Participants) | 11 | 10
units on a scale
  Change from baseline to 1 month | -2.5 (4.0) | 2.0 (5.9)
  Change from baseline to 3 months (n=11, 9) | -1.8 (4.2) | 1.1 (3.8)
Statistical Analysis 1: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 1 month; Test type: Superiority or Other; p = 0.051, t-test, 2 sided
Statistical Analysis 2: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 3 months; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

3. Secondary Outcome: Change in International Consultation on Incontinence Questionnaire - Short Form Score (ICIQ-SF)
Description: The ICIQ-SF provides a brief and robust measure to assess the impact of symptoms of incontinence on quality of life and outcome of treatment. The questionnaire has 4 items and the score can range from 0 to 21, with greater values indicating increased severity of symptoms and lower quality of life.
Time Frame: baseline, 1 month, 3 months
Population: Analysis was done according to the principle of intention-to-treat. The sample size was reduced to 9 in the DSMO instillation arm at 3 months due to withdrawal for reasons unrelated to study (cancer).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Number analyzed (Participants) | 11 | 10
units on a scale
  Change from baseline to 1 month | -2.4 (5.8) | -0.5 (4.4)
  Change from baseline to 3 months (n=11, 9) | -2.5 (5.1) | 0.8 (4.5)
Statistical Analysis 1: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 1 month; Test type: Superiority or Other; p = 0.42, t-test, 2 sided
Statistical Analysis 2: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 3 months; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

4. Secondary Outcome: Change in Urogenital Distress Inventory (UDI-6)
Description: The UDI-6 measures the effect of urinary incontinence on quality of life. It consists of 6 items, each with the response scale from "0=Not at all" to "3=Greatly." The scores can range from 0 to 18; a low score indicates less impact of incontinence on quality of life.
Time Frame: baseline, 1 month, 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Number analyzed (Participants) | 11 | 10
units on a scale
  Change from baseline to 1 month | -1.9 (3.7) | -0.1 (1.9)
  Change from baseline to 3 months (n=11, 9) | -0.9 (3.6) | -0.4 (3.5)
Statistical Analysis 1: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 1 month; Test type: Superiority or Other; p = 0.18, t-test, 2 sided
Statistical Analysis 2: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 3 months; Test type: Superiority or Other; p = 0.77, t-test, 2 sided

5. Secondary Outcome: Number of Participants With Decrease in Blaivas-Groutz Anti-Incontinence Score at 1 Month and 3 Months
Description: The Blaivas-Groutz Anti-incontinence scale was used as a measure of urinary incontinence. This scale combines information on the number of incontinent episodes in a 24-hour period, 24-hour pad weights, and a qualitative rating by the patient into a single score ranging from 0 to 6. this score is then used to categorize incontinence as none (0), mild (1-2), moderate (3-4), or severe (5-6).
Time Frame: baseline, 1 month, 3 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Number analyzed (Participants) | 11 | 10
participants
  1 month | 6 | 4
  3 months (n=11, 9) | 6 | 2
Statistical Analysis 1: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to one month; Test type: Superiority or Other; p = 0.67, t-test, 2 sided
Statistical Analysis 2: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change from baseline to 3 months; Test type: Superiority or Other; p = 0.20, t-test, 2 sided

6. Secondary Outcome: Number of Participants With a Decrease in Urinary Urgency at 1 Month and 3 Months
Description: Urinary urgency was measured by the Indevus Urgency Severity Scale (IUSS). The IUSS asks patients to assess the severity of 'urgency' at each void. The scale employs the following wording: "Degree of urgency is meant to describe your urge to urinate. Sometimes you may feel a very strong urge to urinate and at other times, you may feel a milder urge prior to the onset of a toilet void. Rate this feeling by circling 0, 1, 2, or 3, defined as: 0: NONE - no urgency, 1: MILD - awareness of urgency, but it is easily tolerated and you can continue with your usual activity or tasks, 2: MODERATE - enough urgency discomfort that it interferes with or shortens your usual activity or tasks, 3: SEVERE - extreme urgency discomfort that abruptly stops all activity or tasks."
Time Frame: Baseline, 1 month, 3 months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Number analyzed (Participants) | 11 | 10
participants
  1 month | 4 | 1
  3 months (n=11, 9) | 5 | 0
Statistical Analysis 1: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change between baseline and one month; Test type: Superiority or Other; p = 0.31, t-test, 2 sided
Statistical Analysis 2: Comparison: Botox and DMSO Instillation vs DMSO Instillation; Change between baseline and 3 months; Test type: Superiority or Other; p = 0.038, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Botox and DMSO Instillation | DMSO Instillation
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/10
Other Adverse Events (participants affected / at risk) | 6/11 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox and DMSO Instillation (N=11) | DMSO Instillation (N=10)
Hospitalization for body jerking and termons due to oligodendroglioma. (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization for joint pain due to infection (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization for tibial ulcer (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox and DMSO Instillation (N=11) | DMSO Instillation (N=10)
Urinary Tract Infection (Infections and infestations) | 3 (4) | 5 (6)
High Blood Pressue (Cardiac disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Had fall, unable to walk (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder spasms after instillation (Renal and urinary disorders) | 0 (0) | 1 (1)
Swollen ankles (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nose Bleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Left Distal Radius Fracture from a Twist and Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No